CLINICAL TRIAL: NCT04540107
Title: Metabolic Imaging of Patients With Lower Grade Glioma Using Hyperpolarized 13C Pyruvate
Brief Title: Serial MR Imaging and MR Spectroscopic Imaging for the Characterization of Lower Grade Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Susan Chang (Other)
Collaborators: GE Healthcare (Industry); Sigma-Aldrich (Unknown); Phillips-Medisize (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Susan Chang, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 161016; NCI-2019-08761 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA262630 (NIH); P50CA097257-22 (NIH)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Recurrent World Health Organization (WHO) Grade II Glioma; Recurrent WHO Grade III Glioma; WHO Grade II Glioma; WHO Grade III Glioma
Keywords: Glioma; Hyperpolarized Pyruvate (13C)
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (MRI, MRSI) (CLOSED TO ENROLLMENT) (Experimental): Patients undergo MRI and MRSI scans over 1 hour at baseline. Patients then continue to undergo MRSI scans that follow the clinical MRI schedule set by doctors to monitor patients' care. Participants enrolled in cohort 1 may later enroll in cohort 2 of study once eligibility has been reviewed and approved by neuro-oncologist
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging
- Cohort 2 (MRI, hyperpolarized carbon C 13 pyruvate, MRSI) (Experimental): Patients undergo MRI scan at baseline. Patients then receive hyperpolarized carbon C 13 pyruvate IV over less than 1 minute and undergo MRSI scan at baseline. Patients then continue to undergo MRSI scans that follow the clinical MRI schedule set by doctors to monitor patients' care.
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
  Arms: Cohort 2 (MRI, hyperpolarized carbon C 13 pyruvate, MRSI)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This trial studies how well serial magnetic resonance (MR) imaging and MR spectroscopic imaging work in characterizing lower grade glioma. Diagnostic procedures, such as MR imaging and MR spectroscopic imaging, may detect serial changes in lower grade glioma. This study may help researchers learn more about practical ways of evaluating and standardizing treatment in patients with brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of hyperpolarized 13C MR metabolic imaging as a new and unique tool for making an early assessment of progression and evaluation of response to therapy in patients with lower grade glioma II. To determine whether changes in levels of hyperpolarized 13C pyruvate, lactate and bicarbonate may provide early evidence of tumor progression in patients with lower grade glioma who are being followed with surveillance scans.

III. To determine whether patients with lower grade glioma who are receiving treatment exhibit a reduction in levels of hyperpolarized 13C lactate/pyruvate at follow-up compared to their baseline scan.

OUTLINE: Patients will be enrolled into Cohort 2. Participants previously enrolled in Cohort 1 may enroll in Cohort 2 of study upon re-review of eligibility.

COHORT 1 (CLOSED TO ENROLLMENT): Patients undergo MR imaging (MRI) and MR spectroscopic imaging (MRSI) scans over 1 hour at baseline. Patients then continue to undergo MRSI scans that follow the clinical MRI schedule set by doctors to monitor patients' care.

COHORT 2: Patients undergo MRI scan at baseline. Patients then receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over less than 1 minute and undergo MRSI scan at baseline. Patients then continue to undergo MRSI scans that follow the clinical MRI schedule set by doctors to monitor patients' care.

ELIGIBILITY:
Inclusion Criteria:

* For patients in cohort 1: histologically proven lower grade glioma who are being followed with surveillance scans
* For patients in cohort 2: histologically proven glioma who are scheduled for treatment due to suspected residual or recurrent tumor
* Patients with a life expectancy > 12 weeks
* Patients must have a Karnofsky performance status of >= 60
* Patients must have adequate renal function (creatinine < 1.5 mg/dL) before imaging. These tests must be performed within 60 days prior to the hyperpolarized imaging scan.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to participate in this study or any disease that will obscure toxicity or dangerously impact response to the imaging agent.
* Patients must not have New York Heart Association (NYHA) grade II or greater congestive heart failure
* Patients must not have history of myocardial infarction or unstable angina within 12 months prior to study enrollment
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. Minorities will actively be recruited to participate. No exclusion to this study will be based on race
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must sign an authorization for the release of their protected health information
* Patients may not be known to be human immunodeficiency virus (HIV)-positive. HIV testing is not required for study participation
* Patients must not have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless they are in complete remission and have been off all therapy for that disease for a minimum of 3 years
* Patients must not be pregnant or breast-feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of hyperpolarized imaging scan. Effective contraception (men and women) must be used in subjects of child-bearing potential

Exclusion Criteria:

* Subjects will be excluded from participating in this study if they are unable to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (AEs) | Up to 4 years
  Safety evaluation for endpoint will include monitoring for the occurrence of treatment-emergent adverse events (AEs). Reported toxicities will be graded using the National Cancer Institute (NCI) Common Terminology (Toxicity) Criteria for Adverse Events (CTCAE) version 4.0. All available safety data will be used and will be analyzed using descriptive statistics.
Peak lactate/pyruvate | Up to 4 years
  The peak lactate/pyruvate in tumor and normal appearing brain tissue will be reported.
Peak bicarbonate/pyruvate | Up to 4 years
  The peak bicarbonate/pyruvate in tumor and normal appearing brain tissue will be reported.
Change in peak lactate/pyruvate between scans | Baseline up to 4 years
  The change in peak lactate/pyruvate between scans will be reported.
Change in peak bicarbonate/pyruvate between scans | Baseline up to 4 years
  The change in peak bicarbonate/pyruvate between scans will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04540107/ICF_000.pdf